CLINICAL TRIAL: NCT06390930
Title: Investigating the Effects of Acute Intermittent Hypoxia on Neuroplasticity in Persons With Multiple Sclerosis
Brief Title: Effects of Acute Intermittent Hypoxia on Neuroplasticity in MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00221436
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: multiple sclerosis; plasticity; neuroplasticity; motoneuron; aih; hypoxia; Acute Intermittent Hypoxia; arm; upper extremity
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Hypoxia | interventions — Insemination, Artificial, Homologous

STUDY DESIGN:
Intervention Model Description: randomized, blinded, placebo-controlled, cross-over with repeated measures
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIH first (Experimental): Participants in the first arm will undergo 2 sessions of AIH each separated by a 1-week washout period. 1 week later, participants will undergo 2 sessions of Sham AIH also separated by a 1-week washout period.
  Interventions: Other: Acute Intermittent Hypoxia; Other: Sham Acute Intermittent Hypoxia
- Sham First (Experimental): Participants in the this arm will undergo 2 sessions of Sham AIH each separated by a 1-week washout period. 1 week later, participants will undergo 2 sessions of AIH also separated by a 1-week washout period.
  Interventions: Other: Acute Intermittent Hypoxia; Other: Sham Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — During AIH, the participant will be equipped with a non-rebreathing face mask, and provided with the AIH intervention. The AIH intervention involves alternating breathing cycles. One cycle involves breathing air with lower oxygen concentration (9-10% oxygen) for 30 and 90 seconds, followed by breathing normal room air (21% oxygen) for a similar duration. This cycle is repeated 15 times in one session. Blood oxygen and heart rate are monitored throughout.
  Other Names: AIH
Other: Sham Acute Intermittent Hypoxia — During Sham AIH, the participant will be equipped with a non-rebreathing face mask, and provided with the AIH intervention. The Sham AIH intervention involves alternating breathing cycles. One cycle involves breathing air closely resembling room air (~21% oxygen) for 30 and 90 seconds, followed by breathing normal room air (21% oxygen) for a similar duration. This cycle is repeated 15 times in one session. Blood oxygen and heart rate are monitored throughout.
  Other Names: Sham AIH

SUMMARY:
This study seeks to explore changes in the neural pathways and arm function following a breathing intervention in the multiple sclerosis (MS) population. The breathing intervention, known as Acute Intermittent Hypoxia (AIH), involves breathing brief bouts of low levels of oxygen. Research has found AIH to be a safe and effective intervention resulting in increased ankle strength in people with MS. Here, the study examines arm and hand function before and after AIH. In order to better understand the brain and spinal cord response to AIH, the investigators will measure muscle response, and signals sent from the brain to the arm muscles before and after AIH.

DETAILED DESCRIPTION:
While AIH has shown potential in enhancing neuroplasticity in people with spinal cord injury (SCI), it has yet to be studied extensively in MS. Preliminary research in the MS population demonstrates that a single session of AIH enhances motor output, increasing voluntary muscle strength by as much as 15-20% within 60 minutes. This study will explore potential mechanisms of AIH in MS using measurements of arm function, as well as examination of corticospinal and spinal motoneuron excitability.

Over the past decade, studies have found that brief episodes of modest oxygen reduction (termed AIH) can rapidly enhance neural plasticity in persons with incomplete SCI. AIH activates the serotonergic pathway, leading to increased activity of serotonin receptors and the synthesis of plasticity-related proteins. This plasticity is manifested by a rapid increase in voluntary muscle strength, emerging within 60-90 minutes, in both lower- and upper-limb muscles. The actions of AIH appear to be biologically linked to systems designed to preserve breathing systems that are impaired by damage to the central nervous system (CNS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting MS according to the McDonald criteria, over 5 years ago
* Relapse free for at least 6 months
* Expanded Disability Status Scale (EDSS) ≤7
* Index finger abduction strength <5 according to Medical Research Council Scale, or 9-Hole Peg Test score >20 seconds in at least one hand
* Stable disease modifying therapies for at least 6 months
* Individuals taking dalfampridine will be eligible if taking the same daily dose for at least 2 months prior to screening

Exclusion Criteria:

* Another diagnosis (e.g., peripheral neuropathies or orthopedic) affecting upper limb function
* Mini-Mental State Examination (MMSE) score <24
* Modified Ashworth Scale score >3 on elbow joint
* Uncontrolled hypertension or hypotension (outside 140/90 and 85/55 mmHg)
* History of epilepsy, chronic obstructive pulmonary disease, or sleep apnea
* Unstable medical conditions, ongoing upper limb therapy, or musculoskeletal pain
* Pregnancy as confirmed by urine test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potentials (MEPs) in First Dorsal Interosseous (FDI) | Immediately before, immediately after, and 60 minutes after the intervention.
  The MEPs will be elicited by Transcranial Magnetic Stimulation (TMS), a procedure that uses magnetic fields to stimulate nerve cells in the brain.
Changes in Spinal Reflex Threshold | Immediately before the intervention and immediately after the intervention.
  Spinal reflect threshold will be measured by calculating the average change in threshold length recorded from the biceps tendon's indentation. A linear motor will be used to impose precise tendon indentations of the biceps brachii.
Threshold For Detecting Passive Joint Movement | Immediately before the intervention and immediately after the intervention.
  An assisted movement with enhanced sensation (AMES) will be used to rotate the participant's joint. The difference between the reference and matching joint angles is used to measure joint position sense. The investigators will present three target positions, and subjects will perform ipsilateral matching for each target 5 times.
Accuracy of Direction Estimation of Passive Joint Movement | Immediately before the intervention and immediately after the intervention.
  An AMES will be used to rotate the participant's joint. The difference between the reference and matching joint angles is used to measure joint position sense. The investigators will present three target positions, and subjects will perform ipsilateral matching for each target 5 times.

SECONDARY OUTCOMES:
Grip Strength | Immediately before the intervention and immediately after the intervention.
  The participant will squeeze a calibrated dynamometer to measure grip strength.
Pinch Strength | Immediately before the intervention and immediately after the intervention.
  The participant will pinch a calibrated pinch gauge to measure pinch strength.
Index Finger Abduction Force | Immediately before the intervention and immediately after the intervention.
  Index finger abduction force will be measured using a load cell. We will also record surface EMG activity from the FDI muscle.
Nine-Hole Peg Test | Immediately before the intervention and immediately after the intervention.
  A dexterity measurement involving placing 9 pegs in corresponding holes. Time to complete is measured.
Symbol Digit Modalities Test | Immediately before the intervention and immediately after the intervention.
  A cognition assessment. Using a key, the participant has 90 seconds to match numbers to given geometric figures.
Box and Block Test | Immediately before the intervention and immediately after the intervention.
  A 60 second dexterity measurement involving translating small wooden blocks from one box to another box separated by a partition.
Modified Ashworth Scale | Immediately before the intervention and immediately after the intervention.
  A grading system is applied to the amount of tone felt during a rapid high velocity stretch. The minimal value is 0, and the maximum value is 4. A higher score indicates a higher degree of spasticity.
Ipsilateral Joint Position Matching Task | Immediately before the intervention and immediately after the intervention.
  The participant's hand will be passively moved to a target joint position and then returned to a base position. Participants are then asked to recreate the target joint angle with the same hand. The difference between the reference and matching joint angles is used to measure joint position sense.
Visual Analog Pain Scale | Immediately before the intervention and immediately after the intervention.
  This is used to measure any changes in pain. It is a one-dimensional scale where the patient marks their pain on a 10-cm ruler. The minimal value is 0, and the maximum value is 10. The higher the score, the greater the pain is.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We do not currently have a plan to share IPD.